CLINICAL TRIAL: NCT04459091
Title: Effects of Supplementation With Amino Essential Acids on Circulating Albumin Levels in Patients With Cerebral Ictus in Rehabilitation Phase
Brief Title: Effects of Supplementation With Amino Essential Acids on Circulating Albumin Levels in Stroke in Rehabilitation Phase
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Collaborators: University of Pavia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 2112
Record Dates: First submitted 2020-06-22; First posted 2020-07-07 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Stroke Rehabilitation
Keywords: Serum Albumin; Essential Amino Acid; Functional Recovery
MeSH Terms: interventions — Amino Acids, Essential

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amino essential acids (Experimental): oral supplementation with a mixture of amino essential acids 8 gr die in two administrations for six weeks
  Interventions: Dietary Supplement: Amino Essential Acid
- Placebo (Placebo Comparator): placebo consisting in isocaloric product containing maltodextrins in two administrations for six weeks
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: Amino Essential Acid — 8 gr die in two administration
  Arms: Amino essential acids
Dietary Supplement: placebo — 8 gr die in two administration
  Arms: Placebo

SUMMARY:
In addition to its physiological functions, serum albumin plays a role of neuroprotection in cerebrovascular stroke. The circulating levels of albumin may be reduced in patients with stroke due to the presence of a systemic inflammatory state and to the inadequacy of protein-energy intake. The circulating levels of albumin have proven to be predictors of functional recovery in ischemic stroke and cerebral hemorrhage.

In the present survey it is hypothesized that it is possible to significantly improve the values of hypoalbuminemia by supplementation with essential amino acids and that, in the second place, any increase in albumin may result in a strengthening of functional recovery in patients with a stroke.

DETAILED DESCRIPTION:
In addition to its physiological functions, serum albumin plays a role of neuroprotection in cerebrovascular stroke. The circulating levels of albumin may be reduced in patients with stroke due to the presence of a systemic inflammatory state and to the inadequacy of protein-energy intake. In the patients admitted to the Montescano Neuromotor Rehabilitation Division, the prevalence of hypoalbuminemia is high at the time of admission and remains high, even if decreased, at discharge. The circulating levels of albumin have proven to be predictors of functional recovery in ischemic stroke and cerebral hemorrhage. In the present survey it is hypothesized that it is possible to significantly improve the values of hypoalbuminemia by supplementation with essential amino acids and that, in the second place, any increase in albumin may result in a strengthening of functional recovery in patients with a stroke.

Several factors induce the use of free essential amino acids: they are the most efficient inducers of protein synthesis and albumin is a protein; free essential amino acids and not those contained in proteins allow a more reliable use of the isoleucine and tryptophan, true nutrients limiting the hepatic synthesis of albumin; the free essential amino acids have a faster and complete intestinal absorption of the essential amino acids derived from protein digestion.

ELIGIBILITY:
Inclusion Criteria:

* first episode of cerebral stroke
* first taken in rehabilitation after hospitalization in the acute department

Exclusion Criteria:

* neoplasia
* long-term corticosteroid therapy (> 3 weeks) in the pre-event period and at the time of admission to the rehabilitation department

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-09-15 (Actual)

PRIMARY OUTCOMES:
Serum Albumin Levels | eight weeks
  Number of patients who at discharge show levels of albuminemia> 0.35 gr / dl (normal level)

SECONDARY OUTCOMES:
Functional Independence Measure | eight weeks
  The Functional Independence Measure (FIM) is an 18-item measurement tool that explores an individual's physical, psychological and social function. The tool is used to assess a patient's level of disability. Range total FIM score 18-126. High score corresponds to better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- ICS Maugeri IRCCS, U.O. di Rieducazione e Recupero Funzionale di Montescano, Montescano, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rodriguez de Turco EB, Belayev L, Liu Y, Busto R, Parkins N, Bazan NG, Ginsberg MD. Systemic fatty acid responses to transient focal cerebral ischemia: influence of neuroprotectant therapy with human albumin. J Neurochem. 2002 Nov;83(3):515-24. doi: 10.1046/j.1471-4159.2002.01121.x. PMID 12390513
- [Background] Kimura Y, Yamada M, Kakehi T, Itagaki A, Tanaka N, Muroh Y. Combination of Low Body Mass Index and Low Serum Albumin Level Leads to Poor Functional Recovery in Stroke Patients. J Stroke Cerebrovasc Dis. 2017 Feb;26(2):448-453. doi: 10.1016/j.jstrokecerebrovasdis.2016.10.008. Epub 2016 Nov 14. PMID 27856112
- [Result] Aquilani R, Maestri R, Boselli M, Achilli MP, Arrigoni N, Bruni M, Dossena M, Verri M, Buonocore D, Pasini E, Barbieri A, Boschi F. The relationship between plasma amino acids and circulating albumin and haemoglobin in postabsorptive stroke patients. PLoS One. 2019 Aug 14;14(8):e0219756. doi: 10.1371/journal.pone.0219756. eCollection 2019. PMID 31412042